CLINICAL TRIAL: NCT01502267
Title: Phase 2 Study of Desensitization Protocol for Highly Sensitized Wait Listed Patients
Brief Title: Desensitization Protocol for Highly Sensitized Patients on the Waiting List for Kidney Transplant
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11374
Record Dates: First submitted 2011-12-24; First posted 2011-12-30 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: End Stage Renal Disease
Keywords: Waiting list; Deceased donor kidney transplantation; Desensitization; anti HLA antibody
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Immunoglobulins, Intravenous; Rituximab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (No Intervention): This group will not receive IVIG and B cell depleting agents
- Group 2 (Experimental): This group will receive IVIG and B cell depleting agents
  Interventions: Drug: High dose IVIG and B cell depleting agents

INTERVENTIONS:
Drug: High dose IVIG and B cell depleting agents — 1. IVIG(2g/kg two times on day 1, 30)
  2. Rituximab(375mg/m2 on day 3)
  3. Bortezomib(1.3mg/m2 four times on day 31, 34, 38, 41)
  Other Names: IVIG; Mabthera; Velcade
  Arms: Group 2

SUMMARY:
The purpose of this study is to determine whether high dose IVIG and B cell depleting agents can be used effectively in highly sensitized wait-listed patients.

DETAILED DESCRIPTION:
HLA sensitization is known to be the most important barrier to deceased donor kidney allocation. Therefore, the investigators need to develop better strategies for managing pre-sensitized patients using desensitization protocol. In this study the investigators will used two kinds of medication for the reduction of circulating antibodies (high dose IVIg, B cell depleting agents) to highly-sensitized patients who are on the waiting list for a deceased donor kidney transplantation. After desensitization, the investigators will check that this treatment can increase their chances of receiving a kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* patients who are on the waiting list more than 4 years
* PRA I or II > 50%

Exclusion Criteria:

* Recent recipients of any live attenuated vaccine(s) within 4 weeks
* Subjects who have received IVIG or B cell depleting agents previously
* Subjects with positive result for viral hepatitis(B,C) or HIV infection
* Subjects with active infection
* Lactating or pregnant females
* Subjects who have history of malignancy in recent 5years
* Subjects who have experience of treatment for the psychiatric problem in recent 6months
* Subjects who have hematologic abnormality (Hb < 7g/dL, Platelet < 100,000/mm3, AST/ALT > 80IU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2010-01; Primary Completion 2014-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
The rates of kidney transplantation | from one to five years

SECONDARY OUTCOMES:
Reduction in anti-HLA alloantibodies | 1year
Renal allograft survival | from one to five year
  graft and patient survival
The number of serious complication | from one to five year

CONTACTS AND LOCATIONS:
Overall Officials: Curie Ahn, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Jeong JC, Jambaldorj E, Kwon HY, Kim MG, Im HJ, Jeon HJ, In JW, Han M, Koo TY, Chung J, Song EY, Ahn C, Yang J. Desensitization Using Bortezomib and High-dose Immunoglobulin Increases Rate of Deceased Donor Kidney Transplantation. Medicine (Baltimore). 2016 Feb;95(5):e2635. doi: 10.1097/MD.0000000000002635. PMID 26844479